CLINICAL TRIAL: NCT00869089
Title: An Open Label, Single Center Study to Assess the Safety and Efficacy of a 24 Week Treatment Course of CC-10004 in Adults With Recalcitrant Nodularis
Brief Title: Safety and Efficacy of CC-10004 for Prurigo Nodularis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Neil Korman, Principle Investigator, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102652; 12-07-24 (Other: Institutional Review Board (IRB) Number)
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-09

CONDITIONS: Prurigo Nodularis
Keywords: PN
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-10004 (Experimental): CC-10004 treament:
  30mg,oral medication, BID, for 24 weeks (60mg total DAILY)
  Interventions: Drug: CC-10004

INTERVENTIONS:
Drug: CC-10004 — 30mg,oral medication, BID, for 24 weeks (60mg total DAILY)
  Other Names: apremilast

SUMMARY:
This trial will include:

* Study period up to 7 months.
* Office visits monthly lasting approximately 1 hour.
* Blood Draws.
* Oral medication that is taken 2 times daily.
* Photographs and biopsies if agreed.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form
* Must be male or female and aged ≥ 18 years at time of consent
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must have a diagnosis of prurigo nodularis based on clinical and histological findings and have failed four weeks of treatment with topical therapies, including corticosteroids and/or vitamin D derivatives.
* Must meet the following laboratory criteria:

  * Hemoglobin WNL
  * Hematocrit WNL
  * White blood cell (WBC) count WNL
  * Neutrophils ≥ 1500 /dL
  * Platelets ≥ 100,000 /dL
  * Serum creatinine ≤ 1.5 mg/dL
  * Total bilirubin 2.0 mg/dL
  * Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]) 1.5x upper limit of normal (ULN)
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening (Visit Must have a negative purified protein derivative (PPD) within 28 days of the baseline visit.
* Must have a negative purified protein derivative (PPD) within 28 days of the baseline visit.

Exclusion Criteria:

* History of cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major diseases deemed clinically significant by the investigator
* Any systemic treatment (including ultraviolet light, corticosteroids, thalidomide, azathioprine, cyclosporine) within 28 days of study drug administration.
* Any topical treatments (including corticosteroids, vitamin D derivatives) within 14 days of study drug initiation.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Korman, M.D.,PhD., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was open from September 2008 through 2009. Study visits were conducted in outpatient Dermatology clinic.
Pre-assignment Details: This was an open label single site study for adults with recalcitrant prurigo nodularis. Participants must have failed 4 weeks of treatment with topical corticosteroids or vitamin D derivatives.
Groups:
- CC-10004: CC-10004 treatment:
  30mg,oral medication, BID, for 24 weeks (60mg total DAILY)
Period: Overall Study
Arm/Group | CC-10004
Started | 5
Completed | 2
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Screen Fail | 1

BASELINE CHARACTERISTICS:
Population: Number of subjects enrolled in the study.
Groups:
- CC-10004: CC-10004 Treatment
Arm/Group | CC-10004
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  Age < 18 | 0
  Age > or = 18 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Prurigo Nodularis
Time Frame: 24 weeks
Population: Subjects who completed the study were analyzed.
Measure: Number; unit: participants
Arm/Group | CC-10004
Number analyzed (Participants) | 2
participants
  Response to treatment | 0
  Minimal or no response to treatment | 2

ADVERSE EVENTS:
Arm/Group | CC-10004
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CC-10004 (N=5)
Nausea (Gastrointestinal disorders) | 1 (1)
Headaches (General disorders) | 1 (1)
Prurigo Nodularis Flare (Skin and subcutaneous tissue disorders) | 1 (1)
Worsening of peripheral neuropathy (Nervous system disorders) | 1 (1)
Conjunctival hemorrhage (Eye disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
GI upset (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tongue tenderness (General disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No